CLINICAL TRIAL: NCT01437696
Title: How Much Vitamin D is Required to be Protective Against Deficiency During the Winter Months? - An Investigation in Veterans Living at Ste-Anne's Hospital
Brief Title: How Much Vitamin D is Required to be Protective Against Deficiency During the Winter Months?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Hope Weiler, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HW-11-02
Record Dates: First submitted 2011-09-15; First posted 2011-09-21 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Vitamin D Deficiency
Keywords: Aging; Vitamin D; Bone health; Inflammation; Men
MeSH Terms: conditions — Vitamin D Deficiency; Inflammation; Multiple Endocrine Neoplasia Type 1 | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vitamin D fortified food 500 IU (Experimental): One portion of a specific food item will be provided each day. 500 IU Vitamin D added.
  Interventions: Dietary Supplement: Vitamin D
- Vitamin D fortified food 1000 IU (Experimental): One portion of a specific food item will be provided each day. 1000 IU Vitamin D added.
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): One portion of a specific food item will be provided each day. No vitamin D added.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — A liquid cholecalciferol at a dosage of 500IU will be added to a specific food and provided to the participants once a day for 24 weeks.
  Arms: Vitamin D fortified food 500 IU
Dietary Supplement: Vitamin D — A liquid cholecalciferol at a dosage of 1000IU will be added to a specific food and provided to the participants once a day for 24 weeks.
  Arms: Vitamin D fortified food 1000 IU
Other: placebo — No liquid cholecalciferol will be added to the food.
  Arms: Placebo

SUMMARY:
Vitamin D is essential to bone health. In Canada, it is obtained by sunlight exposure of the skin (between April and October) or by a few foods such as fatty fish, eggs or fortified milk and margarine. This study has 3 main goals which are to determine if Veteran's have enough vitamin D stored in their body, if adding a supplement of 2000 IU/d is enough to correct low vitamin D stores and, if specially formulated foods using an approved vitamin D supplement, are appropriate to maintain vitamin D stores in relation with functional and cognitive status. Initially, a 2000 IU supplement of vitamin D will be provided for 8 weeks. After this period, the participants will be randomly separated into 3 groups (Group A, B or C) for a period of 24 weeks. Group A will receive their usual menu. Group B will receive their usual menu with 1 portion of food containing 500 IU of added vitamin D. Group C will receive their usual menu with 1 portion of food containing 1000 IU of added vitamin D. Food intake will be assessed every 8 weeks and blood samples will be taken every 4 weeks to monitor change in blood concentration of vitamin D and other indicators of bone health. The investigators will document weight and height, hand grip strength, the mid-arm and mid-calf circumferences, the capacity to perform activities of daily living, the number of prescriptions and changes in health condition. The investigators will also take an X-ray the tibia and upper arm to document the amount and quality of bones in those regions. A total of 60 veterans of Ste-Anne's Hospital will participate in this study. Knowing more about vitamin D status and intake will help in confirming the required vitamin D recommendations for the elderly men living in long-term care institutions.

DETAILED DESCRIPTION:
The main objectives of the proposed 2 phase-protocol in aged Canadian veterans (n=60) are to evaluate the impact of 2000 IU/day of vitamin D3 supplementation (tablets or liquid form) on correcting low vitamin D status and the associated impact on biochemistry, bone health markers and markers of inflammation in a Fall period (Before and After, 8 weeks) and, 2) evaluate which food-based supplementation will maintain vitamin D3 status thereafter from winter through spring by measuring serum 25(OH)D concentration following intake of vitamin D delivered (with liquid form vitamin D3) using foods as the vehicle providing an additional 1000 IU/day or 500 IU/day compared to regular meals offered at Ste-Anne's Hospital (SAH) (Randomized Controlled Trial, 3 groups, 24 weeks). Anthropometry (weight, height, BMI, mid-arm and mid-calf circumferences), grip strength, biochemical markers of bone health (25(OH)D, PTH, calcium, ionized calcium and phosphate), assessments of cognitive and functional status (Mini-Mental State Evaluation, Frail Elderly Functional Assessment, Physiotherapy Functional Mobility Profile and Pain Assessment Checklist) as well as volumetric bone mineral density using peripheral quantitative computed tomography (pQCT) will be gathered.

The long-term goal of the research program is to use novel food-delivery systems and approaches to enhancing vitamin D intake that meets the needs of this population. For years, medications have been delivered through foods but few studies have applied this to natural health products such as vitamin D. In chronic care, the number of prescription pills is high often 13 or more not accounting for multiple administrations over a day. Further documentation of health related indicators such as capacity to perform daily activities and chronic pain intensity would relate to quality of life and improve our understanding of vitamin D in more than bone health related issues. The reality of long-term care facilities (financial, human and material resources) needs to be addressed for the newly developed delivery modes to meet the needs of these residents and the projected increase in care required for our aging Canadian population. Large scale interventions will need to take place to give more insight on efficacy and efficiency of this new food delivery approach.

ELIGIBILITY:
Inclusion Criteria:

* All Veterans over the age of 70 years will be invited to participate given selection and exclusion criteria. Level 1, 2 and 3 care will comprise the recruitment pool. These levels of care permit such investigation and do not include those in palliative conditions.
* Individuals with chronic diseases will be permitted to participate as long as the disease is not end-stage (ie prognosis of more than 4 months).
* Not excluding co-morbidities or poor cognition is consistent with the work of others in the area.
* Lastly combined oral and enteral feeding modes will be included since the majority quickly transition to foods but some do take a meal-replacement/liquid supplement.

Exclusion Criteria:

* End-stage renal disease due to altered vitamin D metabolism and use of vitamin D analogues
* End-stage liver disease
* Untreated hyperparathyroid conditions such as cancer and metabolic bone disease except for osteoporosis and osteomalacia
* Any condition that requires enteral feeding alone as feeding route will be excluded since this oral intake, even if only partial, is a critical measurement.

Min Age: 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in 25(OH)D plasma concentrations | Baseline and following 8 weeks of the observation phase. Also following 1, 2, 3, 4, 5 and 6 months of the active supplementation phase.
  Fasted morning blood samples will be taken monthly for assessment of 25(OH)D plasma concentrations.
Changes in Vitamin D intake from foods and supplements | Baseline and following 8 weeks of the observation phase. Also following 2, 4 and 6 months of the active supplementation phase.
  Using food records, vitamin intake will be assessed for 3 days. The records will be collected by a registered dietitian.

SECONDARY OUTCOMES:
Change in bone mineral density | Baseline and following 6 months of the active supplementation phase (32 week timepoint).
  Using peripheral quantitative computed tomography (pQCT) bone mineral density will be assessed for the radius and tibia.
Changes in functional mobility | Baseline and following 32 weeks of study involvement
  Functional mobility will be assessed using grip strength, frail elderly functional assessment (FEFA) and physiotherapy functional mobility profile (PFMP). The assessments will be conducted by the doctoral student and a physiotherapist.
Change in chronic pain over time | Baseline and following 8 weeks of the observation phase. Also following 6 months of the active supplementation phase (32 week timepoint).
  Chronic pain will be assessed using PACSLAC: Pain Assessment Checklist for Seniors with Limited Ability to Communicate.
Changes in biochemistry measurements during the study period | Baseline and following 8 weeks of the observation phase. Also following 2, 4 and 6 months of the active supplementation phase.
  Fasted morning blood sample will be taken to assess calcium, ionized calcium, phosphate, glucose, sodium, potassium, albumin, hemoglobin, and total protein.
Changes in inflammatory markers and bone metabolism markers | Baseline and following 8 weeks of the observation phase. Also following 2, 4 and 6 months of the active supplementation phase.
  Fasted morning blood sample will be taken to assess inflammatory markers: CRP, IL-6, IL-12, IL-14, and TNF alpha. Bone metabolism will be assessed by CTX and osteocalcin.
Change in PTH | Baseline and following 8 weeks of the observation phase. Also following 1, 2, 3, 4, 5 and 6 months of the active supplementation phase.
  Fasted morning blood samples will be taken monthly for assessment of PTH plasma concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Hope A Weiler, PhD, RD, Principal Investigator — McGill University
Locations (1):
- Ste. Anne's Hospital, Ste. Anne-de-Bellevue, Quebec, Canada